CLINICAL TRIAL: NCT02275728
Title: Evaluating the Effectiveness of Pelvic Floor Muscle Training With and Without EMG Biofeedback and Quality of Life in Peri and Postmenopausal Women With Stress Urinary Incontinence.
Brief Title: Pelvic Floor Muscle Training With and Without Biofeedback in Women With Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Adriane Bertotto, Maria Celeste Osório Wender, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02605013.9.0000.5327; 14-0233 (Other: Comitê de Ética Hospital de Clínicas)
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Menopause; Urinary Incontinence, Stress
Keywords: Menopause; Stress Urinary Incontinence; EMG Biofeedback; Pelvic Floor Muscle Training; Quality of life; Physical Therapie
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pelvic Floor Muscle Training(PFMT) (Experimental): The conducted training by two groups, consisting of phasic contractions (3 sets of 10 repetitions of maximal contraction for two seconds to double or triple rest), endurance (two sets of six repetitions of sustained contractions of 6-10 seconds with the same rest time) and training effort, requesting the anticipated contraction of the abdominal pelvic floor coughing effort. We used the same protocol in the supine position, sitting and standing, as evolution of the patient. Both were treated 2 times per week, 20 minutes, totaling 8 sessions.
  Interventions: Other: Pelvic floor muscle training
- EMG Biofeedback treatment (Active Comparator): In this group, the same protocol of the TMAP will be held, however, emg biofeedback is used during training for 20 minutes, 2 times a week, 8 sessions.
  Interventions: Other: Pelvic floor muscle training; Other: Eletromyography Biofeedback
- no treatment (No Intervention): In this group, will be held only the initial assessment, you will not receive treatment for a month and will be reevaluated after being serviced this period.

INTERVENTIONS:
Other: Pelvic floor muscle training — assessment and intervention group with a training of the pelvic floor muscles, another group with training of the pelvic floor muscles and electromyographic biofeedback and a control group will be held. All groups respond to a questionnaire of quality of life. At the end, all groups will be reassessed and compare the effectiveness of interventions between groups.
  Arms: EMG Biofeedback treatment; Pelvic Floor Muscle Training(PFMT)
Other: Eletromyography Biofeedback
  Arms: EMG Biofeedback treatment

SUMMARY:
This study evaluates the action of the pelvic floor muscle training with and without EMG Biofeddback in the treatment of stress urinary incontinence in menopausal, peri and post menopausal women and their quality of life before and after the interventions.

DETAILED DESCRIPTION:
The Pelvic floor muscle training has been the first line of choice in the treatment of Stress Urinary Incontinence. The goal of this technique is increasing the strength and function of the pelvic floor which aims to support the pelvic viscera, as well as part of their duties, such as locks sphincter muscles.

Risk factors such as advanced age, obesity, multiple pregnancy, can cause a woman to present urinary incontinence (SUI), where the main cause is the dysfunction of the pelvic floor muscles and the lack of awareness of these muscles as well as biomechanical problems.

Some studies describe the use of EMG biofeedback to assess and improve the function of the pelvic floor muscles, however, the studies are not yet conclusive about the action of adding this equipment in the treatment of SUI.

In this regard, the EMG Biofeedback has the ability to physiologically evaluate these disorders and perform a faster treatment for these patients, improving their quality of life. The EMG has the ability to monitor and measure the progression of activation of the pelvic floor muscles, giving feedback to the patient and therapist about the actual condition of muscle function.

ELIGIBILITY:
Inclusion Criteria:

Will be included in this study:

* all women,
* spontaneous free will,
* have knowledge of research and sign the Instrument of Consent -TCLE.
* Menopausal women,
* pre and post-menopause,
* urinary incontinence with the effort

Exclusion Criteria:

Will be excluded from the study:

* patients with neurological, cardiovascular, rheumatologic diseases,
* diabetes mellitus,
* chronic lung disease,
* rheumatoid arthritis,
* Enhlers-danlos,
* Sexually Transmitted Diseases (STDs),
* do not submit annual gynecological exams.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pelvic floor muscle strength with "Oxford Scale" | 1 month
  The evaluation consists in bidigital intravaginal test which evaluates the pelvic floor muscle strength using the following 0-5 scale, where 0 = no contraction and 5 = maximal contraction with support against gravity The graduates range from 0 - 5 = 0 has no muscle contraction, 1 = outline of muscle contraction, 2 = contracts without support against gravity, 3 = contracts and holds little against gravity, 4 = contracts and holds up to 6 seconds against gravity and 5 = contracts and holds more than 6 seconds against gravity ntravaginal bidigital test that evaluates scale of pelvic floor muscle strength.
  The graduates range from 0 - 5 = 0 has no muscle contraction, 1 = outline of muscle contraction, 2 = contracts without support against gravity, 3 = contracts and holds little against gravity, 4 = contracts and holds up to 6 seconds against gravity and 5 = contracts and holds more than 6 seconds against gravity

SECONDARY OUTCOMES:
The myoelectric activity evaluation of the pelvic floor | 1month
  The myoelectric activity evaluation of the pelvic floor [Time Frame: 1month] [Safety Issue: No] assessment of myoelectric record by EMG biofeedback through an intra-cavity disposable electrode which evaluates the initial and final rest in 60 seconds, the average of three maximal voluntary contractions, time of sustained contraction, number of peaks of contraction in 10 seconds and the test effort requesting cough

OTHER OUTCOMES:
Measuring quality of life throughInternational Consultation on Incontinence Questionnaire | 1 month
  Is a brief instrument, translated into Portuguese, presents its psychometric properties such as validity, reliability and responsiveness previously tested, consists of three questions related to frequency, severity of urinary loss and its impact on QoL. Presents a range of eight items assess the possible causes or situations of urinary loss. The ICIQ score (ICIQ E) is the sum of scores for questions three, four and five and ranges from 0 to 21 The impact on QoL is defined according to the score of question 5: (0)

CONTACTS AND LOCATIONS:
Overall Officials: Adriane Bertotto, Principal Investigator — Federal University of Rio Grande do Sul

REFERENCES:
- [Result] Kaya S, Akbayrak T, Gursen C, Beksac S. Short-term effect of adding pelvic floor muscle training to bladder training for female urinary incontinence: a randomized controlled trial. Int Urogynecol J. 2015 Feb;26(2):285-93. doi: 10.1007/s00192-014-2517-4. Epub 2014 Sep 30. PMID 25266357
- [Result] Ayeleke RO, Hay-Smith EJ, Omar MI. Pelvic floor muscle training added to another active treatment versus the same active treatment alone for urinary incontinence in women. Cochrane Database Syst Rev. 2013 Nov 20;(11):CD010551. doi: 10.1002/14651858.CD010551.pub2. PMID 24259154
- [Result] Dannecker C, Wolf V, Raab R, Hepp H, Anthuber C. EMG-biofeedback assisted pelvic floor muscle training is an effective therapy of stress urinary or mixed incontinence: a 7-year experience with 390 patients. Arch Gynecol Obstet. 2005 Dec;273(2):93-7. doi: 10.1007/s00404-005-0011-4. Epub 2005 Jul 6. PMID 16001201